CLINICAL TRIAL: NCT06135935
Title: Postprandial Glycaemic Changes When Patients With Type 2 Diabetes Consume the New KDD Products
Brief Title: Postprandial Glucose Response Using Mass-Market No-Added-Sugar Ice Cream
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, CMO, Dasman Diabetes Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: RA HM 2023-002
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; no added sugar-flavored ice cream; conventional ice cream; postprandial glycemic response
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: In this double blind randomized controlled cross over design trial, patients will be randomized to receiving new KDD product or analog first. On the subsequent visit the opposite product will be provided.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-added-sugar ice cream (Experimental): KDD is developing a new line of no-added-sugar products in line with its metabolic reengineering initiative and its metabolic matrix. Four new flavored milks and four new ice creams all have no added sugar. Flavors include chocolate, vanilla, strawberry, and banana. The recipes fundamentally do not alter total saturated fat or protein levels and mainly offer the benefit of no added sugar and a significant reduction in net carbohydrates as well glycemic index.
  Interventions: Other: No-added-sugar ice cream
- conventional products (Active Comparator): KDD has been a leading manufacturer of food and beverages with added sugar (conventional products). The majority of people with type 2 diabetes consume their food products.
  Interventions: Other: Conventional products

INTERVENTIONS:
Other: No-added-sugar ice cream — The initial focus of this clinical trial will be the impact on postprandial glycaemia of 300g of ice cream, since, from a nutrition perspective, the flavored milks and ice creams are very similar in composition.
  Arms: No-added-sugar ice cream
Other: Conventional products — The overconsumption of sugar-added conventional products leads to an increased risk of poor control of glycaemic levels.
  Arms: conventional products

SUMMARY:
KDD is developing a new line of no-added-sugar products in line with its metabolic reengineering initiative and its metabolic matrix. The recipes fundamentally do not alter total saturated fat or protein levels and mainly offer the benefit of no added sugar and a significant reduction in net carbohydrates as well glycaemic index.

DETAILED DESCRIPTION:
The consumption of highly ultra-processed foods has been identified as having detrimental effects on human metabolic health, leading to various adverse health outcomes. The Metabolic Matrix represents a highly quantified, science-based tool for reengineering products with the aim of promoting positive metabolic outcomes. This approach may also contribute to creating shared value by solving important social problems such as obesity and type 2 diabetes by scalable products that are profitable.

KDD is committed to addressing the pandemic of metabolic diseases in Kuwait and would like to develop products that benefit the collective metabolic health of the Kuwait population. KDD is working with partners to assist in its ground-breaking work and to support its efforts with a strong evidence-base rooted in leading-edge science in metabolic health and nutrition. We hypothesise that no-added sugar-flavored ice cream have a substantially different postprandial glycaemic response compared to conventional products in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. Aged over 18 years
3. HbA1c 6.5-8.5% (48-69 mmol/L)

Exclusion Criteria:

1. Lactose intolerant
2. Not liking chocolate ice cream

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-12 (Actual); Primary Completion 2023-12-12 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be area under curve for the plasma glucose response over 120 minutes after consumption of the ice creams. | 8 months
  The aim of this study is to test the postprandial glycemic response after consuming the new no added sugar-flavored ice cream compared to conventional products in patients with type 2 diabetes.

SECONDARY OUTCOMES:
Plasma insulin responses over 120 minutes after consumption of the ice creams. | 8 months
CGM monitor readouts over 24 hours after consumption of the ice creams. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ebaa Al Ozairi, MD, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Ebaa Al Ozairi, Kuwait City, Dasman, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Al-Ozairi E, Mandani Y, Alfaleh G, Raj J, Alshammari S, Le Roux CW. Reformulating ice cream to improve postprandial glucose response: an opportunity for industry to create shared value. Front Nutr. 2024 Jul 16;11:1349392. doi: 10.3389/fnut.2024.1349392. eCollection 2024. PMID 39081682